CLINICAL TRIAL: NCT05092100
Title: Neural Mechanisms for Reducing Interference During Episodic Memory Formation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06302015.045
Record Dates: First submitted 2021-09-15; First posted 2021-10-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Behavior
Keywords: behavior, memory
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Behavioral (Experimental): This arm will use behavioral procedures to test memory for different visual stimulus conditions.
  Interventions: Behavioral: Visual stimulus similarity
- fMRI pattern similarity (Experimental): This arm will use fMRI and behavioral methods to test memory for different visual stimulus conditions.
  Interventions: Behavioral: Visual stimulus similarity; Other: fMRI
- eye tracking (Experimental): This arm will use eye tracking and behavioral methods to test memory for different visual stimulus conditions.
  Interventions: Behavioral: Visual stimulus similarity; Behavioral: Eye tracking

INTERVENTIONS:
Behavioral: Visual stimulus similarity — Visual stimulus similarity will be varied in order to test for effects on memory. Learning protocol (the order and frequency with which stimuli are learned) will also be varied.
  Other Names: Learning protocol
Other: fMRI — fMRI will be used to measure patterns of BOLD activity during learning.
  Arms: fMRI pattern similarity
Behavioral: Eye tracking — Eye tracking will be used to measure patterns of eye movements when viewing images.
  Arms: eye tracking

SUMMARY:
Healthy individuals from the University of Oregon and surrounding community will be recruited for participation in behavioral, fMRI and eye tracking experiments that investigate human memory. Recruitment will involve emails, flyers, and local advertisements. Individuals between the ages of 18-80 (or 18-35 for some studies) will be eligible.

The broad objective of the research is to understand how humans form distinct memories for similar experiences. Experimental sessions will involve studying and trying to remember various images (e.g., images of natural scenes). The intervention will involve manipulating the similarity and/or learning protocol for the studied images. Outcome measures will include (a) behavioral measures of memory, and/or (b) fMRI measures of hemodynamic activity, and/or (c) eye tracking measures of gaze direction. Experimental sessions will last approximately 1-3 hours.

DETAILED DESCRIPTION:
Objective: The goal of the research studies is to understand how memories are formed for similar experiences such that interference (confusion) between these memories is minimized. Of particular interest is the role of the hippocampus (a brain region important for memory).

Participants: Healthy individuals from the University of Oregon and surrounding community will be recruited through fliers, emails, and advertisements. For some of the studies, individuals between 18-80 years of age will be recruited. For others, individuals between 18-35 will be recruited.

Design: All studies will involve studying and trying to remember various images (e.g., natural scenes) displayed on a computer screen. Memory decisions will be made and recorded using a computer keyboard or external button box. The similarity of images and/or the specific learning procedures (e.g., number of repetitions, order of study, etc.) will be manipulated. Experimental sessions will be conducted in behavioral testing rooms (with or without eye tracking equipment) and/or in an MRI scanner.

Outcomes: Measures of interest will include (a) behavioral responses, (b) fMRI measures of hemodynamic responses, and/or (c) gaze direction as measured by eye tracking equipment. Behavioral responses will consist of simple memory decisions, such as indicating whether or not an image has been seen before or trying to remember associations between images. fMRI data will be analyzed using multivariate pattern similarity analyses. Eye tracking data will be used to measure the specific spatial locations of images that participants fixate on.

ELIGIBILITY:
Inclusion Criteria:

Participants in behavioral studies must be:

* healthy and between the ages of 18-35 years old
* native English speakers
* right-handed.

Participants in fMRI studies must be:

* healthy and between the ages of 18-80 years old
* native English speakers
* right-handed.

Exclusion Criteria:

For behavioral studies:

- Potential participants will be informed that use of psychoactive drugs, mental health disorders, and chronic or temporary sleep deficits (an average of less than 6 hours of sleep over the past month or less than 4 hours of sleep the night prior to the experimental session) are reasons for exclusion because of the potential influence on cognitive functioning.

For fMRI studies:

* For some sub-studies, individuals older than age 35 will be excluded because of potential differences in cognitive and brain function across age groups that are beyond the scope of the proposed studies.
* Individuals will be informed that use of psychoactive drugs, mental health disorders, and chronic or temporary sleep deficits (an average of less than 6 hours of sleep over the past month or less than 4 hours of sleep the night prior to the experimental session) are reasons for exclusion because of the potential influence on cognitive functioning.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 737 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Behavior | Data will be collected over a 5 year period. Results from sub-studies will be analyzed within 6 months of the conclusion of data collection.
  Behavioral responses will be recorded by keyboard or external button boxes. These responses will be used to assess the accuracy with which participants remember individual images. Accuracy will be averaged across stimuli within each learning condition to obtain measures of mean memory accuracy (i.e., the percentage of stimuli that were successfully remembered) per condition and participant.
fMRI pattern similarity | Data will be collected over a 5 year period. Results from sub-studies will be analyzed within 6 months of the conclusion of data collection.
  fMRI will be used to measure hemodynamic (BOLD) responses as participants study images. Pattern similarity analyses will be applied to the fMRI data. Pattern similarity will be indexed by the correlation (r) between patterns of BOLD activity. Pattern similarity will be computed for images within and across different learning conditions.
eye tracking | Data will be collected over a 5 year period. Results from sub-studies will be analyzed within 6 months of the conclusion of data collection.
  Eye tracking equipment will be used to measure gaze direction and fixations as participants study images. These data will be used to calculate variables such as the number of saccades (eye movements) made and the percentage of time (within each trial) spent looking at each portion of an image. Data from individual trials will be averaged across trials within each learning condition. This will yield mean values per condition and participant.

CONTACTS AND LOCATIONS:
Overall Officials: Brice A Kuhl, Ph.D., Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified fMRI data will be shared via a public repository
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be made available approximately at the time of (or before) manuscript publication. At the latest, data will be made available 1 year after manuscript publication.
Access Criteria: Data will be publicly accessible.